CLINICAL TRIAL: NCT03553277
Title: Spatial Repellent Products for Control of Vector-borne Diseases - Dengue
Brief Title: Spatial Repellents for Arbovirus Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18-01-4370
Record Dates: First submitted 2018-01-23; First posted 2018-06-12 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Arbovirus Infections
Keywords: Dengue; Zika; Chikungunya; Spatial repellent; transfluthrin
MeSH Terms: conditions — Arbovirus Infections; Dengue; Zika Virus Infection; Chikungunya Fever | interventions — transfluthrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfluthrin (Experimental): transfluthrin
  Interventions: Other: transfluthrin
- Placebo (Placebo Comparator): inert ingredients
  Interventions: Other: placebo

INTERVENTIONS:
Other: transfluthrin — passive emanator with formulated transfluthrin
  Arms: Transfluthrin
Other: placebo — passive emanator with formulated inert ingredients
  Arms: Placebo

SUMMARY:
Dengue viruses are the most medically important arthropod-borne pathogens worldwide, with transmission occurring in most tropical and sub-tropical regions. An estimated 390 million infections occur yearly. Although, there are considerable ongoing efforts to develop a vaccine, vector control remains the only option for reducing dengue virus (DENV) transmission and disease burden. The recent emergence of Aedes-borne Zika (ZIKV) and Chikungunya viruses (CHIKV) highlight need for novel vector control tools. The goal of this project is to determine the efficacy of a spatial repellent (SR) product (active ingredient transfluthrin) for reducing contact between household residents and vector mosquitos and as a result reduce DENV, ZIKV, and/or other Aedes-borne virus transmission. Henceforth the investigators will designate the combined risk of Aedes-borne dengue, Chikungunya, Zika virus transmission by (DCZV). Spatial repellency is used here as a general term to refer to a range of insect behaviors caused by airborne chemicals that reduce contact between people and disease vectors. This can include movement away from a chemical stimulus, and interference with host detection (attraction-inhibition) and/or feeding response.

DETAILED DESCRIPTION:
Protection provided by this product will be measured using entomological and virological approaches, comparing entomological indices will be measured through standard household monitoring of Aedes aegypti population densities, while DCZV transmission will be measured through door-to-door surveillance for active dengue disease and through serological monitoring for DCZV exposure in a randomized cluster trial.

The investigators will establish a cohort of 3,400 persons, primarily children 2-12 years of age and adults who have not been previously infected with DCZV who will provide annual blood samples when they are healthy (longitudinal cohort), whereas in the same clusters the investigators expect to monitor up to 27,500 residents for active dengue disease (febrile surveillance cohort). The cohort will be monitored for a period of 2 years. The use of spatial repellents has never been tested on a large scale to reduce disease and could change vector control practices worldwide, reducing the amount of chemical insecticides applied and also prevent the development of insecticide resistance. The investigators plan to implement a short questionnaire to determine levels of acceptability and perceived efficacy amongst participating households.

The project will be carried out in the Amazonia City of Iquitos, Peru, which has a well-established infrastructure for studying urban dengue fever. The study will generate rigorous evidence, documenting and evaluating the impact of SR products on human infection rates, to be considered and used by academia, industry and public health key stakeholders at the global, regional, national and/or local level and drive efforts to acquire full recommendation of SR products for inclusion in disease control programs.

ELIGIBILITY:
LONGITUDINAL SEROCONVERSION Individual Level

Inclusion Criteria:

* ≥ 2 years of age
* plans to stay in study area for minimum of 12 months
* resident of household or frequent visitor (~20% of day hours in house/mo)

Exclusion Criteria:

* < 2 years of age
* temporary visitor to household
* plans to leave study area within next 12 months

FEBRILE SURVEILLANCE Household Level

Inclusion Criteria:

* adult head of households agree to health visits and census
* individuals spend a minimum of 4hrs per week during the daytime hours or sleep in the house. Temporary residents can be included.

Exclusion Criteria:

* households where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile)
* sites where no residents spend time during the day (i.e., work 7d a week outside the home)

FEBRILE SURVEILLANCE Individual Level

Inclusion Criteria:

* individual who spends a minimum of 4 hours per week within the household
* ≥ 2 years of age
* fever at the time of presentation or report of feverishness within the previous 24 hours or presenting with a rash, arthralgia, arthritis or non-purulent conjunctivitis (suspicion of Zika determined by project physician)

Exclusion Criteria:

* <2 years of age
* individuals who have spent less than 4 hours in the household during the week prior to illness

ENTOMOLOGICAL MONITORING Household Level

Inclusion Criteria:

* adult head of households agrees to survey

Exclusion Criteria:

* properties where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile)

SPATIAL REPELLENT INTERVENTION Household Level

Inclusion Criteria:

* adult head of households agrees to intervention deployment and to provide access to team member at 2-3 week intervals to change product

Exclusion Criteria:

* properties where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile)

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18240 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Aedes-borne virus (ABV) infection. | 2 years
  Compare laboratory confirmed Aedes-borne dengue, Zika virus seroconversion rates in subjects residing in households with active and placebo product, receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator for ABV infections.

SECONDARY OUTCOMES:
Clinically apparent laboratory confirmed cases of Aedes-borne virus (ABV) disease. | 2 years
  Compare laboratory confirmed Aedes-borne dengue, Zika virus infection rates in subjects residing in households with active and placebo product, receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator for ABV disease.
Adult female Aedes aegypti indoor abundance. | 2 years
  Compare adult female Aedes aegypti indoor abundance in households with active and placebo product as an indicator for reduced mosquito house entry due to effect of product.
Adult female Aedes aegypti blood fed abundance. | 2 years
  Compare adult female Aedes aegypti blood fed abundance in households with active and placebo product as an indicator for reduced mosquito human contact due to effect of product.
Adult female Aedes aegypti parity rate. | 2 years
  Compare adult female Aedes aegypti parity rates in households with active and placebo product as an indicator for reduced mosquito survival due to effect of product.
Perception of product efficacy. | 2 years
  Compare perceived efficacy of the product to reduce mosquito nuisance in households with active and placebo product as an indicator for product acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Iquitos, Peru